CLINICAL TRIAL: NCT07005869
Title: Brachial Plexus Tumors; Pathological Types and Surgical Approaches: Multi Center Experience
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fadwa Ahmwd Ahmed, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Brachial plexus Tumors
Record Dates: First submitted 2025-05-21; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Brachial Plexus Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- brachial plexus tumors patients (Other): patients who has brachial plexus tumors
  Interventions: Procedure: brachial plexus tumors excision

INTERVENTIONS:
Procedure: brachial plexus tumors excision — excision of brachial plexus tumors

SUMMARY:
Brachial plexus tumors, are rare, present significant challenges due to their intricate anatomical location and potential impact on upper limb function. These tumors arise from nerve sheath cells, including either benign schwannomas and neurofibromas, or as malignant peripheral nerve sheath tumors (MPNSTs), which require early diagnosis and intervention to improve patient outcomes (1). Surgical resection remains the primary treatment modality, aiming to alleviate symptoms and prevent further neurological compromise.

DETAILED DESCRIPTION:
Brachial plexus tumors, are rare, present significant challenges due to their intricate anatomical location and potential impact on upper limb function. These tumors arise from nerve sheath cells, including either benign schwannomas and neurofibromas, or as malignant peripheral nerve sheath tumors (MPNSTs), which require early diagnosis and intervention to improve patient outcomes (1). Surgical resection remains the primary treatment modality, aiming to alleviate symptoms and prevent further neurological compromise.

The choice of surgical approach is influenced by the tumor's size, location, and relationship with surrounding neurovascular structures. Anterior approaches, including supraclavicular and infraclavicular incisions, provide excellent exposure for lesions in the upper and middle parts of the plexus, whereas posterior approaches are preferred for deep-seated or retroclavicular tumors (2). Intraoperative neurophysiological monitoring (IONM) has significantly improved surgical precision, reducing the risk of postoperative deficit .

Advancements in microsurgical techniques, such as nerve grafting and nerve transfers, have improved functional recovery in patients undergoing brachial plexus tumor resection. Early intervention and meticulous dissection help preserve nerve function and minimize postoperative deficits (3). Minimally invasive techniques, including endoscopic and robotic-assisted approaches, are being explored to reduce morbidity and improve surgical precision (4).

Despite progress in surgical management, challenges remain, particularly in cases of malignant tumors where complete resection may not be feasible. Adjuvant therapies, including radiation and chemotherapy, are increasingly utilized for malignant brachial plexus tumors to enhance local control and reduce recurrence rates (5). Long-term follow-up and rehabilitation play a crucial role in optimizing functional recovery, emphasizing the need for a multidisciplinary approach (6).

This review aims to analyze the indications, techniques, and outcomes of different surgical approaches for brachial plexus tumors, providing insights into optimizing patient outcomes while minimizing surgical morbidity.

ELIGIBILITY:
Inclusion Criteria:

.Patients diagnosed with brachial plexus tumors confirmed through imaging

.Age of Patients: Any age .

.patients who are fit for surgery .

Exclusion Criteria:

. Patients with non-tumorous brachial plexus pathologies (e.g., trauma, inflammation).

.Patients with incomplete medical records or lost follow-up data.

.Patients with recurrent tumors previously treated.

.Patients who are unfit for surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
1-motor power and sensory improvment | 2 years
  Clinical:
  Better outcome according to MRC Muscle Power Scale and Numeric Sensory Scale (NSS) The Medical Research Council (MRC) Muscle Power Scale is commonly used to assess motor power in patients. It ranges from 0 to 5, evaluating voluntary muscle contraction against gravity and resistance.
  The Numeric Sensory Scale (NSS) is a simple and effective tool used to assess sensory function.
  It is based on a numerical rating system from 0 to 10, where patients self-report their level of sensation. This scale is commonly used in neurological examinations to evaluate sensory deficits.
Radiological out come | 2 years
  Radiological :
  Postoperative MRI to detect the residual or recurrence of lesions

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ab khallaf, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No